CLINICAL TRIAL: NCT05310539
Title: Rehabilitation Treatment and Early Recovery After "Wedge Resection" for Pulmonary Metastasis Secondary to Bone Cancer: an Observational Study.
Brief Title: Early Recovery After "Wedge Resection" Surgery to Remove Lung Mestastasis Secondary to Bone Cancer.
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: WEDGE
Record Dates: First submitted 2022-03-14; First posted 2022-04-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Metastasis Lung; Bone Neoplasm
Keywords: pulmonary rehabilitation; wedge resection; early recovery
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of the early recovery after wedge resection surgery — To assess the early recovery will be used 1 minute sit to stand, Numeric Rating scale to assess pain, incentive spirometer to assess vital capacity, Borg modified scale to assess dyspnea.

SUMMARY:
After "wedge resection" surgery, the physiotherapy programs proposed in the literature are heterogeneous and there are few data on the outcomes of such treatments in an oncological population for bone cancer.

The aim of the study is to describe the early rehabilitation process after wedge resection surgery secondary to bone tumor pulmonary mestasasis, highlightining the possible functional recovery in the short and medium term after surgery and indentifying the possible prognostic factors.

DETAILED DESCRIPTION:
In Italy, the incidence of primary bone tumors is around 0.8-1 case per 100,000 inhabitants, therefore an estimated 500 new cases of primary malignant bone tumors are estimated each year, affecting more frequently in children and young people. The presence of pulmonary metastasis occurs in 30% of the population with bone cancer and is the most common site of metastasis. Where possible, the elective treatment of lung metastases is ablative surgery and the wedge resection technique is also commonly used in the event of repeated metastasis over time. Pulmonary wedge resection surgery does not follow the anatomical limits of the lung but it is customized according to the metastatic area to be removed, thus differentiating itself from lobectomies and other thoracotomy surgical techniques.

The trend of vital capacity (CV) and forced expiratory volume in 1s (FEV1), after wedge resection surgery, significantly decrease at 3 months compared to the preoperative evaluation, while at 12 months the CV returns to values close to the preoperative ones and FEV1 remains significantly lower. Rehabilitation treatment is part of the multidisciplinary approach for this type of patient in order to prevent post-surgical respiratory complications (PPC) and shoulder girdle dysfunctions, in the treatment of pain and in the recovery of respiratory volumes. Several authors, describing the physiotherapy treatment techniques, include breathing exercises (Active Cycle Breathing Techniques), early mobilization exercises for the lower limbs and the use of volume incentives. The physiotherapy treatment programs proposed in the literature are heterogeneous and there are no data on the feasibility of such treatments in an oncological population for bone cancer.

Patients are enrolled consecutively in a ward of an italian hospital specialized in bone tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* over 12 years of age
* ablative thoracic surgery for metastases localized to the lung and / or chest wall for primary bone cancer
* must be able to perform the "one minute sit-to-stand" test in the preoperative physiotherapy evaluation

Exclusion Criteria:

* ablative thoracic surgery for a diagnosis DIFFERENT FROM that of lung metastases

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients admitted to the ward with a diagnosis of pulmonary metastases from bone cancer will be enrolled consecutively for the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
1 minute sit to stand (Sixth day after surgery) | Sixth day after surgery
  The test requires the person to stand up from a chair, without the help of the arms, fully extending their knees, and sit down the greatest number of times in the time of one minute.

SECONDARY OUTCOMES:
1 minute sit to stand (daily) | every day after surgery up to 7 day; at 3, 6 and 12 months after surgery.
  The test requires the person to stand up from a chair, without the help of the arms, fully extending their knees, and sit down the greatest number of times in the time of one minute.
pain intensity | every day after surgery up to 7 day, twice a day
  numeric rating scale (from 0 (no pain) to 10 (worst possible pain))
vital capacity (ml) | every day after surgery up to 7 day, twice a day
  the vital capacity will be assess with incentive spirometer named "respirex"
heart rate (bpm) | once a day, before and after 1 minute sit to stand test, up to 7 day
  beats per minute; it will be assess with pulse oximeter
peripheral oxygen saturation (SpO2 %) | once a day, before and after 1 minute sit to stand test, up to 7 day
  it will be assess with pulse oximeter
mBorg Score | once a day, before and after 1 minute sit to stand test, up to 7 day
  dyspnea (shortness of breath, sometimes described as "air hunger") it will be assess using Borg Modified Scale, from 0 to 10, when 0 means "none" (better outcome) and 10 means "maximum" (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: marco cotti, pt, Principal Investigator — IOR - Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vijayamurugan N, Bakhshi S. Review of management issues in relapsed osteosarcoma. Expert Rev Anticancer Ther. 2014 Feb;14(2):151-61. doi: 10.1586/14737140.2014.863453. Epub 2013 Nov 26. PMID 24308680
- [Background] Mori S, Shibazaki T, Noda Y, Kato D, Nakada T, Asano H, Matsudaira H, Ohtsuka T. Recovery of pulmonary function after lung wedge resection. J Thorac Dis. 2019 Sep;11(9):3738-3745. doi: 10.21037/jtd.2019.09.32. PMID 31656646
- [Background] Bohannon RW, Crouch R. 1-Minute Sit-to-Stand Test: SYSTEMATIC REVIEW OF PROCEDURES, PERFORMANCE, AND CLINIMETRIC PROPERTIES. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):2-8. doi: 10.1097/HCR.0000000000000336. PMID 30489442
- [Background] Vaidya T, de Bisschop C, Beaumont M, Ouksel H, Jean V, Dessables F, Chambellan A. Is the 1-minute sit-to-stand test a good tool for the evaluation of the impact of pulmonary rehabilitation? Determination of the minimal important difference in COPD. Int J Chron Obstruct Pulmon Dis. 2016 Oct 19;11:2609-2616. doi: 10.2147/COPD.S115439. eCollection 2016. PMID 27799759
- [Background] Tremblay Labrecque PF, Harvey J, Nadreau E, Maltais F, Dion G, Saey D. Validation and Cardiorespiratory Response of the 1-Min Sit-to-Stand Test in Interstitial Lung Disease. Med Sci Sports Exerc. 2020 Dec;52(12):2508-2514. doi: 10.1249/MSS.0000000000002423. PMID 32555023
- [Background] Kohlbrenner D, Benden C, Radtke T. The 1-Minute Sit-to-Stand Test in Lung Transplant Candidates: An Alternative to the 6-Minute Walk Test. Respir Care. 2020 Apr;65(4):437-443. doi: 10.4187/respcare.07124. Epub 2019 Oct 22. PMID 31641072
- [Background] Tarrant BJ, Robinson R, Le Maitre C, Poulsen M, Corbett M, Snell G, Thompson BR, Button BM, Holland AE. The Utility of the Sit-to-Stand Test for Inpatients in the Acute Hospital Setting After Lung Transplantation. Phys Ther. 2020 Jul 19;100(7):1217-1228. doi: 10.1093/ptj/pzaa057. PMID 32280975
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Wyser C, Stulz P, Soler M, Tamm M, Muller-Brand J, Habicht J, Perruchoud AP, Bolliger CT. Prospective evaluation of an algorithm for the functional assessment of lung resection candidates. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1450-6. doi: 10.1164/ajrccm.159.5.9809107. PMID 10228110
- [Background] Weiner P, Man A, Weiner M, Rabner M, Waizman J, Magadle R, Zamir D, Greiff Y. The effect of incentive spirometry and inspiratory muscle training on pulmonary function after lung resection. J Thorac Cardiovasc Surg. 1997 Mar;113(3):552-7. doi: 10.1016/S0022-5223(97)70370-2. PMID 9081102
- [Background] Schnapp LM, Cohen NH. Pulse oximetry. Uses and abuses. Chest. 1990 Nov;98(5):1244-50. doi: 10.1378/chest.98.5.1244. PMID 2225973
- [Background] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034